CLINICAL TRIAL: NCT03945149
Title: A Double-blind Placebo-controlled Clinical Trial to Evaluate the Chronic Safety and Tolerance of Turmipure Gold™ in Healthy Subjects
Brief Title: A Clinical Trial to Evaluate the Chronic Safety and Tolerance of Turmipure Gold™ in Healthy Subjects
Acronym: TURBIO-GOLD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Givaudan France Naturals (Industry)
Collaborators: BioFortis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: ID-RCB 2019-A00299-48
Record Dates: First submitted 2019-05-06; First posted 2019-05-10 (Actual); Last update posted 2020-12-24 (Actual); Status verified 2020-12

CONDITIONS: Gastrointestinal Tolerance; Liver Function; Kidney Function

STUDY DESIGN:
Intervention Model Description: This safety and tolerance study is designed as a monocentric, randomized, parallel arms, double-blind, placebo-controlled clinical trial.
  Three visits planned: a screening visit (V0) for subjects selection, a randomization visit (V1 with product dispensation, 2 weeks after V0) and a end-of-study visit (V2, 5 weeks after V1). between V1 and V2, a telephone interview will be organized with each subject to evoke the tolerance of the product at mid-term.
  An additional end-of-study visit could be planned if the biological results of the V2 visit are not satisfactory, according to the opinion of the investigator.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Turmipure Gold™ (Active Comparator): 30 subjects will be randomized under active arm and will receive Active Product at V1 and until V2 (5 weeks of treatment).
  Interventions: Dietary Supplement: Turmipure Gold™
- Placebo (Placebo Comparator): 30 subjects will be randomized under Placebo arm and will receive placebo Product at V1 and until V2 (5 weeks of treatment).
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Turmipure Gold™ — 30 subjects will take 1000mg in 4 capsules (with 250ml water before breakfast , each day, during 5 weeks
  Arms: Turmipure Gold™
Dietary Supplement: Placebo — 30 subjects will take 4 capsules with 250ml water before breakfast , each day, during 5 weeks
  Arms: Placebo

SUMMARY:
The aim of this study is to evaluate the safety and tolerance of Turmipure Gold™ product during a chronic consumption of 5 weeks in healthy subjects. The hypothesis of this study is that there are no alterations of the gastrointestinal tolerance, of the haematological and biochemical profiles due to Turmipure Gold™ consumption compared to placebo.

DETAILED DESCRIPTION:
The rhizome of Curcuma longa (turmeric) is commonly used as a spice and for its medicinal proprieties traditionally in Asian countries. Turmeric has been studying in different therapeutic area. Antioxidant, anti-inflammatory (respiratory system, joints and digestive), antimutagenic, antimicrobial, neurological disease, hepatoprotective and anticancer properties are supported by in vitro and in vivo data.

Despite several data identified in the scientific literature, the community herbal monograph of the European Medicines Agency allows the traditional use only for the following therapeutic indication "Traditional herbal medicinal product used to increase bile flow for the relief of symptoms of indigestion (such as sensation of fullness, flatulence, and slow digestion)." According to the World Health Organization (WHO) Monographs on Selected Medicinal Plants, the use for treatment of acid, flatulent, or atonic dyspepsia is supported by clinical data. Treatment of peptic ulcers, and pain and inflammation due to rheumatoid arthritis and of amenorrhoea, dysmenorrhoea, diarrhoea, epilepsy, pain, and skin diseases are uses described in pharmacopoeias and in traditional systems of medicine.

Several health claims are pending for European Commission's decision (referred to the Regulation n°1924/2006). As a consequence, in European countries, claims related to antioxidant, joints, digestion, liver, etc. are tolerated for the moment.

Curcumin has been studied as the main bioactive component of turmeric associated to the potential health effect. However, besides curcumin, others components have been identified called the curcuminoids groups. Curcuminoids are natural yellow-orange pigments and hydrophobic polyphenols derived from the rhizome of the herb Curcuma longa. They are commonly isolated from the spice and food-coloring agent turmeric. Extracts of curcuminoids generally contain 75-80% curcumin, 15-20% demethoxycurcumin (DMC), and 0-10% bisdemethoxycurcumin (BDMC).

Regarding the intrinsic property, curcuminoids have higher solubility in organic solvents than in water. As a consequence, curcumin has low aqueous solubility and poor gastrointestinal absorption. It was also documented that curcumin have low absorption from the gut, rapid metabolism and rapid systemic elimination. This leads to the conclusion that turmeric has low bioavailability, which limits its use in general health care and as an adjunct in managing various diseases. Indeed, it was found low serum levels and limited tissue distribution irrespective of route of administration. In order to improve the bioavailability of curcumin, several approaches have been undertaken. The use of adjuvant like piperine that interferes with glucuronidation; liposomal curcumin, nanoparticles, phospholipid complex; and structural analogues of curcumin. The tested products are different from technology of bioavailability enhancement. Recently, Naturex has developed a dried emulsion formulation using a turmeric extract mixed together with a quillaja extract, sunflower oil and arabic gum. This formulation is highly dispersible in water and should therefore improve the bioavailability of curcuminoids.

In order to assess the bioavailability of the product Turmipure Gold™, Naturex conducted a clinical study in 2018. The plasmatic concentration profile of total curcuminoids (curcumin, DMC, BDMC and their metabolites) on a 24-hour period after consumption of a single dose of 300 mg Turmipure Gold™ 30% curcuminoids formulation in comparison to the one obtained after consumption of 1500 mg Standard turmeric powder extract 95% curcuminoids was investigated as the primary objective (unpublished yet). A statistical significant difference was observed on the primary outcome which was the dose-normalized Area Under the Curve (AUC) 0-24h of Total curcuminoids. Turmipure Gold™ formulation was significantly higher than Standard turmeric powder extract (adjusted p<0.0001) for this parameter.

Thirty subjects received the products in a cross-over design, 16 women and 14 men and no gender effect was observed on the primary outcome.

Statistical significant differences were also observed on the dose-normalized of Area Under the Cuve (AUC0)-24h of Total curcuminoids between products comparisons: Turmipure Gold™ was higher than Turmeric extract (1500mg) combined with piperine (15mg) or the phytosome formulation (1000mg) (adjusted p<0.0001 for each).

The aim of this double-blind placebo-controlled clinical trial is to evaluate the chronic safety and tolerance of Turmipure Gold™ in healthy subjects during 5 weeks +/- 3 days between visit V1 (dispensation of the product) and visit V2 (normal end-of-study). 60 healthy male and female volunteers with 40/60 ratio will be recruited for this study.

In order to assess the gastrointestinal tolerance, a composite score of gastrointestinal tolerance has been chosen as primary endpoint of the trial. The composite score of GI tolerance will be determined as the sum of the scores of the 4 GI symptoms and the composite score of stool frequency and consistency (score of GI tolerance = bloating score + abdominal cramping score + stomach noises score + flatulence score + stool score).

Regarding the safety concern, the European Medicines Agency (EMA) monograph indicate contraindication for the following pathologies: "Hypersensitivity to the active substance(s), obstruction of bile duct, cholangitis, liver disease, gallstones and any other biliary diseases" (confirmed by the WHO monograph). The only undesirable effect reported are "mild symptoms of dry mouth, flatulence and gastric irritation may occur. The frequency is not known." In addition to this, the safety profile of the comparatives products was assessed good in several published trials. This will be investigated deeper in this trial with all the safety and tolerance parameters. An additional end-of-study visit could be planned if the biological results of the V2 visit are not satisfactory, according to the opinion of the investigator.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 60 years (limits included),
* BMI between 19 and 28kg/m² (limits included),
* Weight stable within ±3kg in the last three months,
* With routine blood chemistry values within the normal range,
* For women: Non menopausal with the same reliable contraception since at least 3 cycles before the beginning of the study and agreeing to keep it during the entire duration of the study (condom with spermicidal gel and estrogen/progestin combination contraception accepted) or menopausal without or with hormone replacement therapy (estrogenic replacement therapy begun from less than 3 months excluded),
* Non-smoking or with tobacco consumption ≤ 5 cigarettes / day and agreeing not to smoke during all experimental sessions (V1 and V2),
* Good general and mental health with in the opinion of the investigator: no clinically significant and relevant abnormalities of medical history or physical examination,
* Able and willing to participate to the study by complying with the protocol procedures as evidenced by his dated and signed informed consent form,
* Affiliated with a social security scheme,
* Agreeing to be registered on the volunteers in biomedical research file.

Exclusion Criteria:

* Suffering from a metabolic or endocrine disorder such as diabetes, uncontrolled or controlled thyroidal trouble or other metabolic disorder,
* Suffering from a severe chronic disease (e.g. cancer, HIV, renal failure, ongoing hepatic or biliary disorders, chronic inflammatory digestive disease, arthritis or other chronic respiratory trouble, etc.) or gastrointestinal disorders found to be inconsistent with the conduct of the study by the investigator (e.g. celiac disease),
* Suffering from liver diseases,
* Current disease states that are contraindicated to subjects with dietary supplementation: chronic diarrhea, constipation or abdominal pain, Inflammatory bowel diseases (Crohn's disease or ulcerative colitis), Cirrhosis, chronic laxatives use…,
* Suffering from Irritable Bowel Syndrome (IBS) diagnosed or not by a medical doctor and treated with chronic medication,
* Having medical history of current pathology which could affect the study results or expose the subject to an additional risk according to the investigator,
* Recent gastroenteritis or food borne illness such as confirmed food poisoning (less than 1 month),
* With a low veinous capital of blood samples according to the investigator's opinion,
* With a known or suspected food allergy or intolerance or hypersensitivity to any of the study products' ingredient (gluten intolerance, celiac disease, etc….),
* Pregnant or lactating women or intending to become pregnant within 3 months ahead,
* Exhibiting alcohol or drug dependence,
* On any chronic drug treatment (for example anticoagulant, antihypertensive treatment, treatment thyroid, asthma treatment, anxiolytic, antidepressant, lipid-lowering treatment, corticosteroids, phlebotonic, venotonic, drug with impact on blood circulation …) excepting oral and local contraceptives,
* Currently taking (and during the last month) any supplementation from botanical origins or with curcumin,
* Currently taking (and during the past 3 months) any prebiotics or probiotics supplementation from food or from dietary supplements,
* With significant change in food habits or in physical activity in the 3 months before the V0 visit or not agreeing to keep them unchanged throughout the study,
* Trying to lose weight with a current or planned in the next 3 months specific diet (hyper or hypocaloric, vegan, vegetarian…) or exercise regimen,
* With a personal history of anorexia nervosa, bulimia or significant eating disorders according to the investigator,
* Consuming more than 3 standard drinks of alcoholic beverage daily for men or 2 daily for women or not agreeing to keep his alcohol consumption habits unchanged throughout the study,
* Having a lifestyle deemed incompatible with the study according to the investigator including high level physical activity (defined as more than 10 hours of significant physical activity a week, walking excluded),
* Taking part in another clinical trial or being in the exclusion period of a previous clinical trial,
* Having received, during the last 12 months, indemnities for clinical trial higher or equal to 4500 Euros,
* Under legal protection (guardianship, wardship) or deprived from his rights following administrative or judicial decision,
* Presenting a psychological or linguistic incapability to sign the informed consent,
* Impossible to contact in case of emergency.

After V0 biological analyses the subject will be considered as non-eligible to the study on the following criteria:

- Control record (Glycaemia, Gamma glutamyl transpeptidase (GGT), ASAT, ALAT, Urea, Creatinine and Complete blood count) with clinically significant abnormality according to the investigator.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2019-05-09 (Actual); Primary Completion 2019-07-26 (Actual); Study Completion 2019-07-26 (Actual)

PRIMARY OUTCOMES:
composite score of gastrointestinal tolerance | 5 weeks +/- 3 days (V2)
  The primary endpoint in this study is the composite score of gastrointestinal tolerance (Bristol stool chart and Lickert scale) after 5 weeks of supplementation +/- 3 days (a.u./day, range 0-50), expressed in a.u
  This composite score will be defined as the sum of the ratings of GI symptoms scores and the composite score of stool frequency and consistency (36):
  Composite GI symptoms tolerance = Bloating score + Abdominal cramping score + Stomach noises score + Flatulence score + Stool score*

SECONDARY OUTCOMES:
Individual gastrointestinal symptoms (Bristol Stool Chart) | V1 (Day 0)
  Bristol Stool chart is used - this scale allows to measure to evaluate stool frequency and consistency. The Bristol Stool Chart or Bristol Stool Scale is a medical aid designed to classify faeces into seven groups. The Bristol Stool Chart shows seven categories of stool:
  Type 1-2 indicate constipation Type 3-4 are ideal stools as they are easier to pass, and Type 5-7 may indicate diarrhoea and urgency.
Individual gastrointestinal symptoms (Bristol Stool Chart) | 5 weeks +/- 3 days (V2)
  Bristol Stool chart is used - this scale allows to measure to evaluate stool frequency and consistency. The Bristol Stool Chart or Bristol Stool Scale is a medical aid designed to classify faeces into seven groups. The Bristol Stool Chart shows seven categories of stool:
  Type 1-2 indicate constipation Type 3-4 are ideal stools as they are easier to pass, and Type 5-7 may indicate diarrhoea and urgency.
Individual gastrointestinal symptoms (Lickert scale) | V1 (Day 0)
  Lickert scale was used to evaluate gastro-intestinal symptoms. The gastro-intestinal symptoms will be reported during 3 days before V1 visit. A mean of these 3 days will be calculated. Each GI symptom will be given a score of 0 (no symptoms) to 10 (severe symptoms).
  This scale allow to have four scores :
  * Bloating score (a.u./day, range 0-10),
  * Abdominal cramping score (a.u./day, range 0-10),
  * Stomach noises score (= Borborygmi) (a.u./day, range 0-10),
  * Flatulence score (a.u./day, range 0-10), These scores will be combined to evaluate the gestointestinal symptoms
Individual gastrointestinal symptoms (Lickert scale) | 5 weeks +/- 3 days (V2)
  Lickert scale was used to evaluate gastro-intestinal symptoms. The gastro-intestinal symptoms will be reported during 3 days before V1 visit. A mean of these 3 days will be calculated. Each GI symptom will be given a score of 0 (no symptoms) to 10 (severe symptoms).
  This scale allow to have four scores :
  * Bloating score (a.u./day, range 0-10),
  * Abdominal cramping score (a.u./day, range 0-10),
  * Stomach noises score (= Borborygmi) (a.u./day, range 0-10),
  * Flatulence score (a.u./day, range 0-10), These scores will be combined to evaluate the gestointestinal symptoms
Haematological safety parameters: blood count-formula | V1 (Day 0)
  blood count-formula
Haematological safety parameters: blood count-formula | 5 weeks +/- 3 days (V2)
  blood count-formula
Sodium mmol/L dosage | V1 (Day 0)
  Biochemical blood safety parameters
Sodium mmol/L dosage | 5 weeks +/- 3 days (V2)
  Biochemical blood safety parameters
Potassium mmol/L dosage | V1 (Day 0)
  Biochemical blood safety parameters
Potassium mmol/L dosage | 5 weeks +/- 3 days (V2)
  Biochemical blood safety parameters
Chloride mmol/L dosage | V1 (Day 0)
  Biochemical blood safety parameters
Chloride mmol/L dosage | 5 weeks +/- 3 days (V2)
  Biochemical blood safety parameters
Calcium mmol/L dosage | V1 (Day 0)
  Biochemical blood safety parameters
Calcium mmol/L dosage | 5 weeks +/- 3 days (V2)
  Biochemical blood safety parameters
Inorganic Phosphorus mmol/L dosage | V1 (Day 0)
  Biochemical blood safety parameters
Inorganic Phosphorus mmol/L dosage | 5 weeks +/- 3 days (V2)
  Biochemical blood safety parameters
Glucose mmol/L or g/L dosage | V1 (Day 0)
  Biochemical blood safety parameters
Glucose mmol/L or g/L dosage | 5 weeks +/- 3 days (V2)
  Biochemical blood safety parameters
Urea mmol/L dosage | V1 (Day 0)
  Biochemical blood safety parameters
Urea mmol/L dosage | 5 weeks +/- 3 days (V2)
  Biochemical blood safety parameters
Creatinine µmol/L dosage | V1 (Day 0)
  Biochemical blood safety parameters
Creatinine µmol/L dosage | 5 weeks +/- 3 days (V2)
  Biochemical blood safety parameters
Total bilirubin µmol/L dosage | V1 (Day 0)
  Biochemical blood safety parameters
Total bilirubin µmol/L dosage | 5 weeks +/- 3 days (V2)
  Biochemical blood safety parameters
Total cholesterol (mmol/L or g/L) dosage | V1 (Day 0)
  Biochemical blood safety parameters
LDL (mmol/L) dosage | V1 (Day 0)
  Biochemical blood safety parameters
LDL (mmol/L) dosage | 5 weeks +/- 3 days (V2)
  Biochemical blood safety parameters
HDL-cholesterol (mmol/L) dosage | V1 (Day 0)
  Biochemical blood safety parameters
HDL-cholesterol (mmol/L) dosage | 5 weeks +/- 3 days (V2)
  Biochemical blood safety parameters
Total cholesterol (mmol/L or g/L) dosage | 5 weeks +/- 3 days (V2)
  Biochemical blood safety parameters
Triglycerides mmol/L or g/L dosage | V1 (Day 0)
  Biochemical blood safety parameters
Triglycerides mmol/L or g/L dosage | 5 weeks +/- 3 days (V2)
  Biochemical blood safety parameters
Alkaline phosphatase (ALP) µkat/L dosage | V1 (Day 0)
  Biochemical blood safety parameters
Alkaline phosphatase (ALP) µkat/L dosage | 5 weeks +/- 3 days (V2)
  Biochemical blood safety parameters
Aspartate aminotransferase (ASAT) µkat/L dosage | V1 (Day 0)
  Biochemical blood safety parameters
Aspartate aminotransferase (ASAT) µkat/L dosage | 5 weeks +/- 3 days (V2)
  Biochemical blood safety parameters
Alanine aminotransferase (ALAT) µkat/L dosage | V1 (Day 0)
  Biochemical blood safety parameters
Alanine aminotransferase (ALAT) µkat/L dosage | 5 weeks +/- 3 days (V2)
  Biochemical blood safety parameters
Total proteins g/L dosage | V1 (Day 0)
  Biochemical blood safety parameters
Total proteins g/L dosage | 5 weeks +/- 3 days (V2)
  Biochemical blood safety parameters
Albumin g/L dosage | V1 (Day 0)
  Biochemical blood safety parameters
Albumin g/L dosage | 5 weeks +/- 3 days (V2)
  Biochemical blood safety parameters
Albumin/globulin ratio. | V1 (Day 0)
  Biochemical blood safety parameters
Albumin/globulin ratio. | 5 weeks +/- 3 days (V2)
  Biochemical blood safety parameters
glucose dosage | V1 (Day 0)
  Urinary safety parameters
glucose dosage | 5 weeks +/- 3 days (V2)
  Urinary safety parameters
protein dosage | V1 (Day 0)
  Urinary safety parameters
protein dosage | 5 weeks +/- 3 days (V2)
  Urinary safety parameters
potential Hydrogen (pH) | V1 (Day 0)
  Urinary safety parameters
potential Hydrogen (pH) | 5 weeks +/- 3 days (V2)
  Urinary safety parameters
blood presence | V1 (Day 0)
  Urinary safety parameters
blood presence | 5 weeks +/- 3 days (V2)
  Urinary safety parameters
ketonic corpse | V1 (Day 0)
  Urinary safety parameters
ketonic corpse | 5 weeks +/- 3 days (V2)
  Urinary safety parameters
nitrites dosage | V1 (Day 0)
  Urinary safety parameters
nitrites dosage | 5 weeks +/- 3 days (V2)
  Urinary safety parameters
density | V1 (Day 0)
  Urinary safety parameters
density | 5 weeks +/- 3 days (V2)
  Urinary safety parameters
bilirubin dosage | V1 (Day 0)
  Urinary safety parameters
bilirubin dosage | 5 weeks +/- 3 days (V2)
  Urinary safety parameters
urobilinogen dosage | V1 (Day 0)
  Urinary safety parameters
urobilinogen dosage | 5 weeks +/- 3 days (V2)
  Urinary safety parameters
leukocytes dosage | V1 (Day 0)
  Urinary safety parameters
leukocytes dosage | 5 weeks +/- 3 days (V2)
  Urinary safety parameters
quality of life score | V1 (Day 0)
  The GastoIntestinal quality of Life (GIQLI) questionnaire is composed of 36 items. The responses for each item are scored from 0 to 4, from the worst to the best rating. Example of answers to question 1: always (0), most of the time (1), sometimes (2), rarely (3), never (4).
  The average overall score for each subject and visit will be calculated by summing the scores of each question divided by 144 and multiplied by 100 (average overall score reduced to a score between 0 and 100; the maximum score being 100) (Slim et al., 1999).
  The items focus on 5 subscales (Slim et al., 1999):
  * Symptoms (19 items): items 1 to 9 and 27 to 36 (theoretical score range: 0-76),
  * Fitness (7 items): items 15 to 21 (theoretical score range : 0-28),
  * Emotions (5 items): items 10 to 14 (theoretical score range: 0-20),
  * Social integration (4 items): items 22, 23, 25 and 26 (theoretical scope range: 0-16),
  * The effect of possible medical treatment (1 item): item 24 (theoretical score range: 0-4).
quality of life score | 5 weeks +/- 3 days (V2)
  The GastoIntestinal quality of Life (GIQLI) questionnaire is composed of 36 items. The responses for each item are scored from 0 to 4, from the worst to the best rating. Example of answers to question 1: always (0), most of the time (1), sometimes (2), rarely (3), never (4).
  The average overall score for each subject and visit will be calculated by summing the scores of each question divided by 144 and multiplied by 100 (average overall score reduced to a score between 0 and 100; the maximum score being 100) (Slim et al., 1999).
  The items focus on 5 subscales (Slim et al., 1999):
  * Symptoms (19 items): items 1 to 9 and 27 to 36 (theoretical score range: 0-76),
  * Fitness (7 items): items 15 to 21 (theoretical score range : 0-28),
  * Emotions (5 items): items 10 to 14 (theoretical score range: 0-20),
  * Social integration (4 items): items 22, 23, 25 and 26 (theoretical scope range: 0-16),
  * The effect of possible medical treatment (1 item): item 24 (theoretical score range: 0-4).
3 days Food diary | V1 (Day 0)
  This diary will be filled by subjects the week before V1 visit and the data will be collected and analyzed by a dietician.
  This diary will allow to evaluate food intake :
  * total energy intake (kcal),
  * percentage of energy intake from proteins (%),
  * percentage of energy intake from fat (%),
  * percentage of energy intake from carbohydrates (%),
  * dietary fiber (g) and hydric intake,
  These data will be combined to evaluate the food intake
3 days Food diary | 5 weeks +/- 3 days (V2)
  This diary will be filled by subjects the week before V2 visit and the data will be collected and analyzed by a dietician.
  This diary will allow to evaluate food intake :
  * total energy intake (kcal),
  * percentage of energy intake from proteins (%),
  * percentage of energy intake from fat (%),
  * percentage of energy intake from carbohydrates (%),
  * dietary fiber (g) and hydric intake,
  These data will be combined to evaluate the food intake
Physical activity global score | V1 (Day 0)
  This self-administered questionnaire IPAQ will be filled by subjects at V1 visit. For each subject and visit, the total metabolic equivalent will be calculated from the IPAQ questionnaire short form.
  This continuous score, expressed as MET-min per week (MET level x Number of minutes of activity/day x Number of days per week), will be calculated using the following formula (Guideline IPAQ, 2005):
  Total MET-minutes/week = Walking (METs*min*days) + Moderate intensity (METs*min*days) + Vigorous intensity (METs*min*days) with: . Walking = 3.3 METs;
  * Moderate Intensity = 4.0 METs;
  * Vigorous Intensity = 8.0 METs.
Physical activity global score | 5 weeks +/- 3 days (V2)
  This self-administered questionnaire IPAQ will be filled by subjects at V2 visit. For each subject and visit, the total metabolic equivalent will be calculated from the IPAQ questionnaire short form.
  This continuous score, expressed as MET-min per week (MET level x Number of minutes of activity/day x Number of days per week), will be calculated using the following formula (Guideline IPAQ, 2005):
  Total MET-minutes/week = Walking (METs*min*days) + Moderate intensity (METs*min*days) + Vigorous intensity (METs*min*days) with: . Walking = 3.3 METs;
  * Moderate Intensity = 4.0 METs;
  * Vigorous Intensity = 8.0 METs

OTHER OUTCOMES:
occurrence of adverse events | V0 (-14days)
  Safety objectives
occurrence of adverse events | V1 (Day 0)
  Safety objectives
occurrence of adverse events | V2 (5 weeks +/- 3 days)
  Safety objectives

CONTACTS AND LOCATIONS:
Overall Officials: Pascale Fança-Berthon, PhD, Study Director — Naturex
Locations (1):
- Biofortis Mérieux NutriSciences, Saint-Herblain, France

IPD SHARING:
Plan to Share IPD: No